CLINICAL TRIAL: NCT02520700
Title: A Comparison of White-light and Daylight Topical Methyl 5-aminolaevulinic Acid Photodynamic Therapy for Actinic Keratoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Dr Paul Collins, Consultant Dermatologist, St Vincent's University Hospital, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2015-07-30; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study participants (Experimental): This was split scalp design - so each patient had one half of scalp treated with daylight PDT and one side treated with the artificial white light PDT - a surgical light (Maquet Power 500 LED surgery light)
  Interventions: Device: Daylight and Maquet Power 500 LED surgery light

INTERVENTIONS:
Device: Daylight and Maquet Power 500 LED surgery light — Comparing the use of daylight and a surgical light (Maquet Power 500 LED surgery light) to activate ALA cream for treatment of actinic keratoses

SUMMARY:
Photodynamic therapy (PDT) uses visible light to treat a premalignant condition, called actinic keratosis, which results on chronically sun exposed skin such as on a balding scalp. A cream is applied containing aminolaevulinic acid or methyl aminolaevulinate and this is converted in the cells to the photodegradable product protoporphyrin IX (PpIX). Visible light causes the degradation of PpIX resulting in the production of reactive oxygen species and then cell death in the actinic keratosis. In conventional PDT a lamp is used to supply the visible light. The main draw back to treatment is pain. Recent studies have shown that daylight can be used as the source of visible light and is as effective as conventional PDT. Patients find this form of treatment less painful and therefore preferable. The reduction in pain seen in daylight PDT appears to be related to the fact that no significant quantity of PpIX accumulates prior to exposure to the light source and small quantities of PpIX are activated continuously during daylight exposure. The drawback of performing daylight PDT in Ireland is the climate, both in terms of cloud cover and temperature. The typical daylight treatment times is 2 hours and it would be difficult for patients to stay outside in winter, spring and autumn. This study investigates the use of an artificial white light source, a Maquet PWD 50SF theatre-light, as an alternative.

DETAILED DESCRIPTION:
Study Summary:

Title:

A Randomized Single-blinded, Prospective Study to compare a Maquet PWD 50SF theatre-light as a light source with natural daylight for the application of photodynamic therapy (PDT) to treat actinic keratoses.

Photodynamic therapy (PDT) is of proven efficacy for treatment of actinic keratosis (AK) and is increasingly used internationally. It involves the topical application of 5-aminolaevulinic acid cream (ALA) or its methyl ester methyl 5-aminolaevulinic acid (MAL), which is absorbed into the AK and converted into a photosensitizing compound protoporphyrin IX. When the AK is then exposed to visible light an oxygen dependent photochemical reaction is induced which results in cell death through apoptosis and necrosis.

Pain is the main limiting factor with PDT. Recently researchers have used natural daylight as the source of visible light for photodynamic therapy, a process called daylight PDT. This has been found to be equally effective as conventional PDT but less painful. Patients prefer this treatment option and in fact in Copenhagen, where they routinely offer daylight PDT from April to October, they have found that patients will frequently opt to defer their treatment until a time of year when daylight PDT is an option. The drawback of performing daylight PDT in Ireland is the climate, both in terms of cloud cover and temperature. The typical daylight treatment time is 2 hours and it would be difficult for patients to stay outside in winter, spring and autumn. This study investigates the use of an artificial white light source as an alternative.

It is not known what is the light dose required to effectively treat AK's, but a study on daylight PDT in Copenhagen found no difference in treatment outcome above 8 J cm-2.

The pain experienced with PDT may relate to the accumulation of PpIX and the short accumulation time of 30 minutes used in daylight PDT may account for some of the reduction in pain experienced with daylight PDT. With PpIX photography it can be demonstrated that with daylight PDT (incubation 30 mins) almost no accumulation of PpIX occurs yet the local reaction (erythema and erosions) and the clinical response indicate that the photodynamic reaction is taking place. Perhaps the key to the tolerability and efficacy of daylight PDT is not allowing so much PpIX to accumulate. The reduction in pain and the efficacy may result from the continuous activation of small quantities of PpIX. It is known from studies looking at PpIX accumulation in psoriasis that PpIX can still be identified in the skin up to 14 days after application of ALA. If the patient spends time outdoors in the days after PDT it is likely that small quantities of PpIX continue to be activated.

Daylight PDT has to date been studied exclusively in Nordic countries and has proved effective, despite the fact that these countries have a relatively low daylight irradiance. Wiegell et al have studied the PpIX light dose at various latitudes between the July and December months. They found that in Copenhagen, Denmark, a country at similar latitude to Ireland (55 degrees north in the former versus 53 degrees north in the later) it was possible to receive a light dose above 8 J cm-2 in 2 hours on nearly every day in July, August and September. In the first three weeks of October this fell to 16 out of 21 days. They also associated the weather conditions with the light dose and in Copenhagen they found that the mean light dose in 2 hours in July and August was 10.6 J cm-2 on rainy days, 30.7 J cm-2 on partly sunny days and 38.3 J cm-2 on sunny days. It was also determined that weekly mean temperatures need to be 10 degrees or higher for a patient to be comfortably treated outdoors. Therefore, patients are treated with daylight PDT in Copenhagen from 20th April to the 24th October.

A large multicenter study of daylight PDT found no difference between 2 hours and 3 hours daylight exposure.

In Copenhagen they perform daylight PDT from April to October and only reschedule the treatment if the day is very rainy and overcast.

The investigators propose to study the use of the Maquet PWD 50SF theatre light as an alternative light source to daylight. This would provide a year-round, well-tolerated treatment option for patients.

The Maquet PWD 500 theatre light source has been chosen for a number of reasons:-

1. It has a suitable spectrum, i.e., it emits radiation in the wave band that reacts most efficiently with the PpIX to give the optimum response,
2. It does not emit UV radiation which this patient subgroup is particularly sensitive to.
3. There is no infrared (IR) radiation emitted which can cause heating and therefore further complications.
4. It has an ideal size and geometry for treating the head.
5. The output and distribution of LEDs is optimal for this application.

Study protocol:

Based on prior studies of similar design, aiming for a significance level of 0.05 and a power of 0.80 and on the assumption that the smallest clinically important mean difference is 15% and the standard deviation of the difference in response is 25%, at least 22 patients need to be enrolled in this study.

The investigators will enrol these patients from the patients who have been referred for PDT. For inclusion patients must be in generally good health and attending for treatment of AKs on the scalp or face. Two symmetrical treatment fields will be defined. AKs in each treatment area will be counted, graded, mapped and photographed. Grading will be according to Olsen et al ; I, mild (more easily felt than seen), II, moderate (easily felt and seen), III, severe (thick obvious AK). Sunscreen with a protection factor of 20 will be applied to all sun exposed areas including the treatment areas (P20; Riemann & Co. A/S, Hilleroed, Denmark). This sunscreen has been chosen to avoid potential absorption of wavelengths activating protoporphyrin IX. In all patients hyperkeratotic lesions will be pre-treated with paraffin gel to remove keratotic debris, carefully avoiding bleeding. No patient will receive pre-treatment analgesia.

All patients will be randomized to determine which side of the scalp is treated first. Randomization will be achieved by the patient choosing an envelope with a card marked right or left. Approximately 1 gram of MAL cream will be applied on the right treatment field. They will then initially have treatment daylight PDT ,weather permitting. The treatment for the second side will be PDT using a Maquet PWD 50SF theatre-light as a light source. After MAL application patients will be instructed to start daylight exposure after 30 minutes or will be positioned below the Maquet PWD 50SF theatre-light. Exposure to daylight or the Maquet PWD light will then be discontinued after 2 hours.

The second treatment field will be treated one week later so that each patient will have daylight PDT to one treatment area and PDT using the Maquet PWD 50SF theatre light as a light source to the other treatment area.

Prior to treatment in both groups fluorescence will be graded on a scale of 1 -3, using a Wood's light; one being light/pale, 2 being moderate and 3 being strong.

For daylight PDT patients will record how long they sat outside and what the weather conditions were like. Any interruption to light exposure must be recorded.

For both treatments patients will rate their pain using a visual analogue score (VAS) (1-100) at 1, 30, 60, 90 and 120 minutes. To use this patients move a counter along a 100 mm scale from "no pain" to "worst pain ever". The flip side of the scale indicates the score numerically. A nurse will record the numerical pain score and patients will not be aware of this value. If treatment has to be discontinued because of pain the timing of this will be recorded. Adverse events will be recorded.

Patient will be reviewed between 1 and 3 days following treatment for adverse events. Patients will be assessed for local reactions such as erythema and erosions and asked to indicate how long pain persisted. To assess clinical response patients will be assessed 28 days after their last treatment. The investigators will record if patients had a preference for one treatment modality. The investigators will use the baseline map and categorize response for AK lesions as complete response or non-complete response. Patients will similarly be assessed at 3 months, 6 months and 9 months for clinical response.

The primary endpoint will be complete response rates of AKs. Secondary endpoints will be pain scores, adverse effects and patient preference.

ELIGIBILITY:
Inclusion Criteria:

* patient requiring treatment for actinic keratoses on forehead or scalp

Exclusion Criteria:

* immunosuppressed patients, those with abnormal photosensitivity, contact allergy to topical therapy for use in the study or pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The reduction in the actinic keratosis count per treatment field | 9 months follow up
  Palpable AKs within those areas defined as treatment fields will be counted, mapped and photographed at baseline and at 1, 3, 6 and 9 months

SECONDARY OUTCOMES:
Pain scores on visual analogue scale (VAS) at 1, 30, 60, 90 and 120 minutes during treatment | 2 hours of treatment duration
Patient satisfaction with treatment, on a scale of zero to ten | At follow up one to three days post treatment
Erythema or erosions (mild/moderate/severe) | 1 - 3 days post treatment
  Patients were clinically assessed 1 - 3 days following each treatment. In each treatment field the degree of erythema was rated by the investigator as mild, moderate or severe. Similarly the presence of erosions was recorded and rated as mild, moderate or severe.

REFERENCES:
- [Derived] O'Gorman SM, Clowry J, Manley M, McCavana J, Gray L, Kavanagh A, Lally A, Collins P. Artificial White Light vs Daylight Photodynamic Therapy for Actinic Keratoses: A Randomized Clinical Trial. JAMA Dermatol. 2016 Jun 1;152(6):638-44. doi: 10.1001/jamadermatol.2015.5436. PMID 26843523